CLINICAL TRIAL: NCT06315374
Title: Exploring the Benefits of a 3D-Printed Aerosolized Medication Delivery Assist Device in Patients With Chronic Respiratory Diseases
Brief Title: 3D-Printed Aerosolized Medication Delivery Assist Device in Patients With Chronic Respiratory Diseases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to persistent challenges in participant recruitment, the study has been terminated and the protocol has been formally withdrawn.
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FJUH112267
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pulmonary Disease
Keywords: Soft mist inhaler; device error; hand strength; finger muscle power; coordination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simply using soft mist inhaler (Active Comparator): Routine use of soft mist inhaler only
  Interventions: Other: Use soft mist inhaler
- Use soft mist inhaler with a 3D assistive device (Experimental): Use soft mist inhaler with a 3D-printed assist device
  Interventions: Device: Use soft mist inhaler with a 3D assistive device

INTERVENTIONS:
Other: Use soft mist inhaler — Only use soft mist inhaler
  Arms: Simply using soft mist inhaler
Device: Use soft mist inhaler with a 3D assistive device — Use soft mist inhaler with a 3D-printed assist device
  Arms: Use soft mist inhaler with a 3D assistive device

SUMMARY:
The purpose of this study is to investigate the auxiliary benefits of three-dimensional printed activating assistive devices for soft-mist inhaler on patients' utilization habit.

DETAILED DESCRIPTION:
Background： The most common treatment for chronic respiratory diseases is inhalation therapy. However, inhalation therapy requires not only correct operating skills, but also exemplary and sustained adherence from the patient. Soft-mist inhaler does not require hand-mouth coordination or minimum inhalation flow rate, and the aerosol release time is longer, which can effectively deliver more medication to the respiratory tract. If the patient is unable to operate the soft-mist inhaler correctly due to abnormal finger joints or weakened hand muscles, it may affect the effectiveness of inhalation.

Study Design： This is a one-year, single-centre, prospective randomized controlled, crossover trial.

Methods： This study will be conducted in the Chest Medicine Education Room on the 2nd floor of Fu Jen Catholic University Hospital. A total of 60 participants will be recruited and randomly assigned into two groups: the control group and the experimental group. Data collection will be conducted after one month of intervention, followed by a crossover trial. Data will be collected again after the second month of intervention, and statistical analysis will be performed.

Effect： This study expect that three-dimensional printed activating assistive devices for soft-mist inhaler will enhance the satisfaction and convenience of elderly patients with chronic respiratory diseases who use soft-mist inhaler, thereby increasing their medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-80 years
* Patients diagnosed with chronic respiratory diseases requiring the use of SMI medication by a physician
* Signed informed consent form

Exclusion Criteria:

* Not a first-time user of SMI medication
* Requires assistance from others (primary caregiver or nurse) for the operation of SMI medication
* Refusal to participate in the trial

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
satisfaction survey | 1 month after the intervention
  feedback and satisfaction regarding the initiation of SMI medication with 3D-printed aerosolized medication delivery assist device (maximun 35 and minimum 7), higher means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan